CLINICAL TRIAL: NCT02852954
Title: Determining Levels of Expression of Progesterone-Induced Blocking Factor in Endometrial Cancer Cells.
Brief Title: Progesterone Induced Blocking Factor Expression Levels in Endometrial Cancer Cells.
Status: Completed | Type: Observational
Sponsor: Kayseri Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erdem Sahin, Director, Kayseri Education and Research Hospital
Other Study IDs: 2016/405
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2016-08

CONDITIONS: Progesterone Induced Blocking Factor in Endometrial Cancer
Keywords: Progesterone Induced Blocking Factor; Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- study group1: 20 paraffin embedded blocks which was diagnosed endometrial cancer
- control group: 20 paraffin embedded blocks of healthy women
- study group2: 20 paraffin embedded blocks which was diagnosed endometrial hyperplasia

SUMMARY:
Immune system suppression effect of Progesterone Induced Blocking Factor(PIBF), it could be questionable whether tumor cells express PIBF for escape of immune system. There are some studies in the literature that evaluate PIBF expression of different malign cells (e.g. glioblastoma multiforme as a malign central nerve system, leukemia, astrocytoma as a primary brain tumor, lung cancer and chorionic carcinoma). According to previous studies PIBF has been used as an anti-tumor immune suppressor by tumor cells. There is no data about the PIBF expression of endometrial tumor cells. Therefore, the investigators aim to determine the PIBF expression levels in the endometrial cancer cells.

DETAILED DESCRIPTION:
This retrospective controlled study will be conducted at both Obstetrics and Gynecology clinics and Pathology clinics of Kayseri Training and Research Hospital. This study will be conducted with the use of formalin fixed paraffin embedded tissue blocks immunohistochemically to determine the PIBF expression levels in the samples. There are three groups in this study; endometrial cancer, endometrial hyperplasia and normal endometrium and each of the groups contained 20 paraffin embedded blocks provided form the Pathology clinic of Kayseri Training and Research Hospital archives.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed endometrial cancer
* diagnosed endometrial hyperplasia

Exclusion Criteria:

* diagnosed cancer except endometrial cancer

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There are three groups in this study; endometrial cancer,endometrial hyperplasia and normal endometrium and each of the groups contained 20 paraffin embedded blocks provided from the Pathology clinic of Kayseri Training and Research Hospital archives.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Immunohistochemically Levels of PIBF in Endometrial Cancer Cells | 3 months